CLINICAL TRIAL: NCT00834405
Title: A Relative Bioavailability, Parallel Study of Leflunomide 20 mg Tablets Under Non-Fasting Conditions
Brief Title: Leflunomide 20 mg Tablets, Non-Fasting
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: B026504
Record Dates: First submitted 2009-01-30; First posted 2009-02-03 (Estimated); Results first posted 2009-08-18 (Estimated); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Leflunomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Leflunomide (Experimental): Leflunomide 20 mg Tablet
  Interventions: Drug: Leflunomide 20 mg Tablets
- Arava® (Active Comparator): Arava® 20 mg Tablet
  Interventions: Drug: ARAVA® 20 mg tablets

INTERVENTIONS:
Drug: ARAVA® 20 mg tablets — 1 x 20 mg, single-dose non-fasting
  Arms: Arava®
Drug: Leflunomide 20 mg Tablets — 1 x 20 mg, single-dose non-fasting
  Arms: Leflunomide

SUMMARY:
The objective of this study is to compare the relative bioavailability of leflunomide 20 mg tablets (manufactured by TEVA Pharmaceutical Industries, Ltd. and distributed by TEVA Pharmaceuticals USA) with that of ARAVA 20 mg tablets (Aventis) in healthy, adult, non-smoking subjects [females (who are unable to become pregnant) and vasectomized males] under non-fasting conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

* All subjects selected for this study will be non-smokers at least 18 years of age. Females must be physically unable to become pregnant. Males must be vasectomized. Weight of the subjects shall not be more than 20% ± from normal for height and body frame (Metropolitan Life, 1993, Height, Weight, Body Chart).
* Each subject shall be given a general physical examination within 21 days of initiation of the study. Such examination includes, but is not limited to, blood pressure, general observations, and history.
* Each female subject will be given a serum pregnancy test as part of the pre-study screening process.
* Adequate blood and urine samples should be obtained within 21 days before beginning of the first period and at th eend of the trial for clinical laboratory measurements.
* Clinical laboratory measurements will include the following:

  1. Hematology: hematocrit, hemoglobin, red blood cell count, platelets, white blood cell count (with differential).
  2. Clinical chemistry: creatinine, BUN, glucose, SGOT/AST, SGPT/ALT, bilirubin, and alkaline phosphatase.
  3. Urine Analysis: pH, specific gravity, protein, glucose, ketones, bilirubin, occult blood, and cells.
  4. HIV Screen: pre-study only.
  5. Hepatitis-B, C Screen: pre-study only.
  6. Drugs of Abuse Screen: pre-study and at check-in before dosing.
* Subjects will be selected if all above are normal.

Exclusion Criteria:

* Subjects with a history of chronic alcohol consumption (during past 2 years), drug addiction, or recent serious gastrointestinal, renal, hepatic or cardiovascular disease, tuberculosis, epilepsy, asthma, diabetes, psychosis or glaucoma will not be eligible for this study.
* Subjects whose clinical laboratory test values are greater than 20% outside the normal range may be retested. if the clinical values are outside the range on retesting, the subject will not be eligible to participate in the study unless the clinical investigator deems the result to not be significant.
* Subjects who have a history of allergic responses to the class of drug being tested should be excluded from the study. Subjects who have a history of allergic responses to cholestyramine should be excluded from the study.
* All subjects will have urine samples assayed for the presence of drugs of abuse as part of the clinical laboratory screening procedures and at check-in before dosing. Subjects found to have urine concentrations of any of the tested drugs will not be allowed to participate.
* Subjects should not have donated blood and/or plasma for at least 30 days prior to the first dosing of the study.
* Subjects who have taken any investigational drug within 30 days prior to the first dosing of the study will not be allowed to participate.
* Female subjects who are pregnant or who are able (women with child bearing potential) to become pregnant during the study will not be allowed to participate.
* All female subjects will be screened for pregnancy at check-in. Subjects with positive or inconclusive results will be withdrawn from the study.
* Male subjects who are physically able to father a child will not be allowed to participate. Male subjects must be vasectomized (at least 3 months) with medical verification.
* Subjects who smoke or use tobacco in any form will not be eligible to participate in the study. Three months abstinence is required.
* Subjects who are unable to tolerate multiple venipuncture will be excluded.
* Subjects who have taken any product containing leflunomide within 180 days of dosing will not be allowed to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2002-04; Primary Completion 2002-05 (Actual); Study Completion 2002-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David B. Erasmus, M.D., Principal Investigator — Cetero Research, San Antonio
Locations (2):
- United States (2):
  - Gateway Medical Research, Inc., Saint Charles, Missouri
  - Bioassay Laboratory, Inc., Houston, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Leflunomide | Arava®
Started | 20 | 17
Completed | 20 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Leflunomide | Arava® | Total
Number analyzed (Participants) | 20 | 17 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 16 | 35
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 23
  Male | 7 | 7 | 14
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 19 | 17 | 36
  Black | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 20 | 17 | 37

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Concentration - Metabolite A77 1726 in Plasma
Description: Bioequivalence based on Cmax
Time Frame: Blood samples collected over 72 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Leflunomide | Arava®
Number analyzed (Participants) | 20 | 17
ng/mL | 2488.000 (385.181) | 2345.294 (266.156)
Statistical Analysis 1: Comparison: Leflunomide vs Arava®; Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-72 and Cmax; Geometric Test/Ref Ratio x 100 = 106, 90% CI [98.0 to 114] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

2. Primary Outcome: AUC0-72 - Area Under the Concentration-time Curve From Time Zero to 72 Hours Post-dose (Per Participant) - Metabolite A77 1726
Description: Bioequivalence based on AUC0-72
Time Frame: Blood samples collected over 72 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Leflunomide | Arava®
Number analyzed (Participants) | 20 | 17
ng*h/mL | 132584.730 (18639.707) | 123335.784 (13732.783)
Statistical Analysis 1: Comparison: Leflunomide vs Arava®; Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-72 and Cmax; Geometric Test/Ref Ratio x 100 = 107, 90% CI [100 to 115] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator is not permitted to discuss or publish trial results.